CLINICAL TRIAL: NCT05606588
Title: Preventing Sensory and Motor Dysfunctions in Children Receiving Neurotoxic Chemotherapy - a Randomized Controlled, Multi-center Trial
Brief Title: Preventing Sensory and Motor Dysfunctions in Children Receiving Neurotoxic Chemotherapy
Acronym: PrepAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Kantonsspital Aarau (Other); Ostschweizer Kinderspital (Other); University Hospital Heidelberg (Other); University Hospital Freiburg (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other); Charite University, Berlin, Germany (Other); National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Fiona Streckmann, Dr., University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-00527
Record Dates: First submitted 2021-05-17; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Pediatric Cancer
Keywords: Cancer; Lymphoma; Leukemia; Non-Hodgkin Lymphoma; Children; Exercise; Chemotherapy-induced peripheral neuropathy; CIPN; Sensorimotor Training
MeSH Terms: conditions — Neoplasms; Lymphoma; Leukemia; Lymphoma, Non-Hodgkin; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will follow a prospective, multicenter, two-armed, randomised, controlled, assessor-blinded trial trial (RCT with follow-up).
Who Masked: Outcomes Assessor
Masking Description: All assessors will be blinded and participants will only be told the result of their randomization after the baseline assessment. For the following assessments patients and guardians will be instructed prior to the assessment not to reveal the arm they are in. Assessors are instructed to converse as little as possible outside the friendly instructions. Assessors and trainers will participate in separate study meetings and cannot speak to each other regarding patient matters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will perform a standardized, age-adjusted, specific playful sensorimotor training (SMT) program twice a week for the duration of their medical therapy, in addition to usual care.
  Interventions: Behavioral: Playful sensorimotor training
- Control group (No Intervention): The control group receives treatment as usual. The control group will be given the opportunity to participate in the intervention after therapy.

INTERVENTIONS:
Behavioral: Playful sensorimotor training — For the max. duration of the first in-hospital phase (3weeks), all children will receive supervised training. When children go home they will be supplied with a manual, specific exercises and the necessary training devices. Regular supervision will allow to ensure that the training is performed at maximum benefit. Each session will last for about 20 to 30 minutes in total, including a child-specific warm-up and cool-down. The children will be asked to maintain balance in a previously acquired "short-foot-position", knees slightly flexed (30°), without shoes. Training will consist of 5 playful balance exercises chosen from a standardized pool of exercises according to the child's age, with increasing difficulty in order to allow for individual, optimal progression. Each of the 5 exercises will contain of 5 repetitions for 10sec. allowing for a 20sec. rest in between each set and a 1min rest between each exercise in order to avoid neural fatigue.
  Arms: Intervention group

SUMMARY:
The investigators would like to conduct a prospective, multicenter, two-armed trial (RCT with follow-up). Patients will be recruited from 7 centers (CH/D). All patients (and their guardians) scheduled to receive chemotherapy containing either a platinum derivate or vinca-alkaloid, will be asked to participate. Willing patients will then be randomized either into an intervention group or a control group. Patients in the intervention group will perform a standardized, age-adjusted, specific playful sensorimotor training (SMT) program twice a week for the duration of their medical therapy, in addition to usual care, while the control group receives treatment as usual. The CG will be given the opportunity to participate in the intervention after therapy. Data will be assessed at 3-4 time points: Prior to chemotherapy (baseline T0), after 12 weeks (T1), after completion of therapy for children that are treated >3 months (Tp) and after 12 months follow-up (T3). Additionally, status of Chemotherapy-induced peripheral neuropathy (CIPN) reported symptoms will be monitored twice in-between (6 weeks).

The investigators hypothesize that less children in the intervention group will develop symptoms of CIPN (TNS score) with its debilitating side-effects. Furthermore, children in the intervention group will be able to maintain relevant motor and sensory functions and their associated physical functions which will enable them to receive their planned medical therapy but also to stay on the age-appropriate motor development level, improve their quality life and enhance social reintegration after therapy.

DETAILED DESCRIPTION:
Modern therapy has improved survival for children with cancer. However, treatment has unintended consequences. Depending on the neurotoxic agent (platinum derivates or vinca-alkaloids), 52%-100% of children develop a peripheral neuropathy. Diagnosis is underreported and its impact as potentially initial cause for many sensory and motor symptoms underestimated. The severe symptoms such as loss of sensation, numbness, pain, absent reflexes as well as loss of balance control not only delays motor development milestones such as walking, running, jumping or climbing, diminishing children's quality of life and affecting their social reintegration, but is also of high clinical relevance. Additionally, recovery is poor and there are currently no effective options to prevent or treat the symptoms of Chemotherapy-induced peripheral neuropathy (CIPN). Promising results have so far been achieved with specific exercise interventions.

The investigators would therefore like to conduct a prospective, multicenter, two-armed trial (RCT with follow-up). Patients N=131 will be recruited from 7 centers: University Children's Hospital of Basel, the Inselspital Bern, Kantonsspital Aarau, Children Hospital for Eastern Switzerland St. Gallen, University Children Hospital Freiburg and the National Center for tumor diseases (NCT), University Children Hospital Heidelberg, Charité Berlin. All patients (and their guardians) scheduled to receive chemotherapy containing either a platinum derivate or vinca-alkaloid, will be asked to participate. Willing patients will then be randomized either into an intervention group or a control group (CG). Patients in the intervention group will perform a standardized, age-adjusted, specific playful sensorimotor training (SMT) program twice a week for the duration of their medical therapy, in addition to usual care, while the control group receives treatment as usual. The CG will be given the opportunity to participate in the intervention after therapy. Data will be assessed at 3-4 time points: Prior to chemotherapy (baseline T0), after 12 weeks (T1), after completion of therapy for children that are treated >3 months (Tp) and after 12 months follow-up (T3). Additionally, status of CIPN reported symptoms will be monitored twice in-between (6 weeks). The investigators hypothesize that less children in the intervention group will develop symptoms of CIPN (TNS score) with its debilitating side-effects. Furthermore, children in the intervention group will be able to maintain relevant motor and sensory functions and their associated physical functions which will enable them to receive their planned medical therapy but also to stay on the age-appropriate motor development level, improve their quality life and enhance social reintegration after therapy.

ELIGIBILITY:
Inclusion Criteria:

* All tumor patients, aged 6-18 years, who are scheduled to receive neurotoxic chemotherapy with a platinum-derivate or vinca- alkaloid (e.g. vincristine, vinblastin mono, carboplatinum, cisplatin).

Exclusion Criteria:

* Exclusion criteria are known neuropathies of other cause (e.g. diabetes), disabilities or lack of German language that prevent the understanding of the informed consent as well as the instructions for training.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 131 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pre-/Post incidence of neuropathic symptoms via Ped-mTNS score | Baseline (T0), subjective screening for symptoms of CIPN (via phone cell), 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 Months (TFU)
  Primary endpoint is the Ped-mTNS score. It contains a short questionnaire as well as a clinical test battery. The questionnaire is composed of three sets of questions on sensory symptoms and pain, motor function, and autonomic function, and a five- part neurologic exam. The clinical test battery contains light touch sensation, evaluated with Semmes-Weinstein-monofilaments, pin sensibility (MediPin), vibration sensibility assessed with a biothesiometer, deep tendon reflexes of Achilles and patellar tendons and muscular strength examined by a manual muscle test36, each category is rated on a likert scale from 0-4 (0 indicating no symptoms and 4 severe symptoms).
Pre/Post change of signs and symptoms of a neuropathy (VAS (0-10)) | Baseline (T0), Screening for symptoms of CIPN (via phone cell), 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 Months (TFU)
  Signs and symptoms of CIPN

SECONDARY OUTCOMES:
Secondary Outcomes - Pre/post change of postural control | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  postural control - sway path on the Leonardo force plate
Pre/post change of Dorsiflexion | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  dorsiflexion function, assessment of foot drop with a goniometer and hand-held dynamometer
Pre/post change of strength in the lower extremity - knee extension | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  knee extension strength will be assessed with a hand-held dynamometer
Pre/post change of lower limb power | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  lower limb power will be assessed with the countermovement jump
Pre/post change of gait speed | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  10m walk test / walk to run transition time
Pre/post change of neuropathic pain | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  CIPN-related pain will be assessed on a child-appropriate visual analogue scale (VAS)
Pre/post change of level of physical activity | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  participation of exercise-related leisure activities
Pre/post change of physical self-concept | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  childrens' physical self concept via questionnaire
Pre/post change of patients' self-reported, health-related quality of life | Baseline (T0), after 12 weeks (T1), within 7days after last dosage of medical therapy (Tp), 12 months after last dose of Chemotherapy (TFU)
  childrens quality of life via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Streckmann, Dr., Principal Investigator — University of Basel, Department of Sport, Exercise and Health
Locations (2):
- Switzerland (2):
  - Kantonspital Aarau, Basel
  - UKBB Kinderspital, Basel

IPD SHARING:
Plan to Share IPD: Yes
data will be shared on request after completion of the study
Supporting Information: Study Protocol
Time Frame: data will be available after completion of the study and publication of the first manuscript
Access Criteria: on demand